CLINICAL TRIAL: NCT04498845
Title: RECLEAN Pilot Study: Reducing Lead in the Homes of Construction Workers
Brief Title: RECLEAN Pilot Study
Acronym: RECLEAN
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Principal invetigator left the institution.
Sponsor: Boston University (Other)
Collaborators: US Department of Housing and Urban Development (U.S. Federal Agency); Centers for Disease Control and Prevention (U.S. Federal Agency); Ohio State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: H-40676; MALTS0013-19 (Other Grant/Funding Number: HUD)
Record Dates: First submitted 2020-07-31; First posted 2020-08-05 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Lead Poisoning
Keywords: Blood lead level; Construction workers; Household member exposure; National Health And Nutrition Examination Survey (NHANES)
MeSH Terms: conditions — Lead Poisoning

STUDY DESIGN:
Intervention Model Description: After a cross sectional preliminary trial of the in-home family educational session in a one time home visit, there will be 3 types of interventions (basic, intermediate, and advanced) conducted in ~20 homes with ~50 participants for each intervention type.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Basic intervention group (Active Comparator): Participants in the basic intervention group will have a 1-hour in-home assessment plan and family educational session.
  Interventions: Other: In-home assessment plan; Behavioral: Family educational session
- Intermediate intervention group (Experimental): Participants in the intermediate intervention group will have a 1-hour in-home assessment plan and educational session and refer worker to a 1-hr worker take home prevention educational session.
  Interventions: Other: In-home assessment plan; Behavioral: Family educational session; Behavioral: Worker take home prevention training
- Advanced intervention group (Experimental): Participants in the advanced intervention group will have a 1-hour in-home assessment plan and educational session, refer worker to a 1-hr worker take home prevention educational session, and provision of D-LEAD all-purpose cleaner and laundry detergent.
  Interventions: Other: In-home assessment plan; Behavioral: Family educational session; Behavioral: Worker take home prevention training; Other: D-LEAD cleaner products

INTERVENTIONS:
Other: In-home assessment plan — The in-home family educational session provides participants with resources to identify and reduce exposures to metals in the home environment.
Behavioral: Family educational session — The 1-hr in-home family educational session, administered during the first home visit to all participants, adapts a motivational interview model to reduce exposure to metals. this done by empowering families to make informed decisions regarding lead and metal exposures in their home environments that originate from different sources with an emphasis on sources from the workplace. The session will consist of both developing a plan tailored for the home and reviewing educational materials on strategies to reduce exposures in the home, focusing on barriers families experience when attempting to change their behaviors.
Behavioral: Worker take home prevention training — The take home prevention 1-hour educational session guides the worker through 6 simple steps to identify and then prioritize change/s that can be made before leaving work to prevent take-home lead. It has been adapted from the AGILE model for prioritizing tasks. Participants will also be provided with a pamphlet about how to prevent lead from being taken home.
  Arms: Advanced intervention group; Intermediate intervention group
Other: D-LEAD cleaner products — D-LEAD cleaner products include hand wipes, all surfaces cleaner and laundry detergent.
  Arms: Advanced intervention group

SUMMARY:
This is an exposure assessment pilot study tailored for families of construction workers living with a child. The investigators will compare home dust metal levels and resident's blood metal levels before and after an educational and environmental intervention. A baseline and a post intervention period assessment will be conducted with home and car lead inspections and risk assessments with collection of dust, urine, blood and toenail samples and a survey.

Objectives of this research are to:

1. To characterize pre-intervention home exposures to lead and other metals in households with one construction worker inhabitant living with a child, by assessing household members' biospecimens and home dust metal levels.
2. To develop and evaluate customized home interventions (including environmental and educational approaches) to reduce metals exposure in three tiers of intervention.
3. To characterize home exposures to lead and other metals post intervention and determine adapted behaviors and whether the degree of metals exposure reduction (including take home exposures) in the households depends on the level of intervention.

ELIGIBILITY:
First, construction workers will be recruited. Second, household members of the construction worker will be recruited.

Inclusion Criteria:

Construction workers must meet all of the following inclusion criteria:

1. 18 years of age or older
2. works full time in construction with high risk for metal exposures
3. lives in the Greater Boston area
4. lives with at least 1 child household member 1 year of age or older (does not have to be a child of the worker but interested in participating in the study)
5. speaks English or Spanish.

Household resident participants must meet all of the following inclusion criteria:

1. child (1 - 17 years of age) or adult (18 years of age or older)
2. lives in the Greater Boston area with the worker participating in this study
3. speaks English or Spanish.

Exclusion Criteria: None

Min Age: 1 Year | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2021-04-27 (Actual); Primary Completion 2024-01-20 (Actual); Study Completion 2024-01-20 (Actual)

PRIMARY OUTCOMES:
Change in lead levels in dust from household wiped surfaces | Baseline, 5 months
  Dust samples will be collected in the home from wiping up to ten 1ft by 1ft surfaces in the home and three wipes in the car following HUD methods from smooth surfaces likely to be contaminated by the worker and that likely expose other family members such as the laundry area, entry walkway, and living room area, as well as areas with potential lead like window sills. Investigators will use SKC 550-002 colorimetric wipe kit for lead on all wipes in order to obtain immediate color response in the presence of lead (reddish color suggests lead). Wipes will be then stored to be sent to the laboratory for quantitative elemental analysis.
Change in lead levels from household vacuumed dust | Baseline, 5 months
  Dust samples will be collected by vacuuming the entire home floors and surfaces into a clean sampling thimble. Participants will be asked not to vacuum the house, if possible, at least one week prior to the scheduled home visit, tso that enough dust is available for testing.
Blood metal levels from adult household members at baseline | Baseline
  During each home visit, a blood sample will be collected from each participant. The frozen blood samples will be sent to the CDC metals laboratory for analysis. Blood will be analyzed using CDC Method for blood multi-element panel, which includes cadmium (Cd), lead (Pb), manganese (Mn), and mercury (Hg).
Blood metal levels from adult household members at 5 months | 5 months
  During each home visit, a blood sample will be collected from each participant. The frozen blood samples will be sent to the CDC metals laboratory for analysis. Blood will be analyzed using CDC Method for blood multi-element panel, which includes cadmium (Cd), lead (Pb), manganese (Mn), and mercury (Hg).
Blood metal levels from child household members at baseline | Baseline
  During each home visit, a blood sample will be collected from each participant. The frozen blood samples will be sent to the CDC metals laboratory for analysis. Blood will be analyzed using CDC Method for blood multi-element panel, which includes cadmium (Cd), lead (Pb), manganese (Mn), and mercury (Hg).
Blood metal levels from child household members at 5 months | 5 months
  During each home visit, a blood sample will be collected from each participant. The frozen blood samples will be sent to the CDC metals laboratory for analysis. Blood will be analyzed using CDC Method for blood multi-element panel, which includes cadmium (Cd), lead (Pb), manganese (Mn), and mercury (Hg).
Blood metal levels from construction workers at baseline | Baseline, 5 months
  During each home visit, a blood sample will be collected from each participant. The frozen blood samples will be sent to the CDC metals laboratory for analysis. Blood will be analyzed using CDC Method for blood multi-element panel, which includes cadmium (Cd), lead (Pb), manganese (Mn), and mercury (Hg).
Blood metal levels from construction workers at 5 months | Baseline, 5 months
  During each home visit, a blood sample will be collected from each participant. The frozen blood samples will be sent to the CDC metals laboratory for analysis. Blood will be analyzed using CDC Method for blood multi-element panel, which includes cadmium (Cd), lead (Pb), manganese (Mn), and mercury (Hg).

SECONDARY OUTCOMES:
Change in household members' knowledge about lead exposure | Baseline, 1 hour after in-home family educational session
  Investigator developed pre- and post-assessments will be administered to participating household members after the in-home family educational session to evaluate their knowledge regarding potential for exposure to lead in their home environment, especially as it relates to the worker's job in construction, and strategies to prevent or reduce that potential for exposure. Higher number of correct answers are associated with greater knowledge.
Change in workers' knowledge about household lead exposure | Baseline, 1 hour after worker educational session
  Investigator developed pre- and post-assessments will be administered to participating workers after the worker educational session to evaluate their knowledge regarding take-home lead exposure, especially as it relates to their job in construction, and strategies to prevent or reduce that potential for exposure. Higher number of correct answers are associated with greater knowledge.
Change in behaviors of household members | 1 month, 5 months
  Self-reported behaviors of household members regarding prevention of lead exposure will be assessed from responses to an investigator developed survey that will be administered after the first and second home visits. The follow-up survey will ask questions on the behavior change of participants since the first home visit and how successfully they have adhered to their home action plan and to describe any challenges they may have faced.

CONTACTS AND LOCATIONS:
Overall Officials: Diana Ceballos Ochoa, PhD, Principal Investigator — BU School of Public Health
Locations (1):
- Boston University School of Public Health, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No